CLINICAL TRIAL: NCT02131012
Title: Intravitreal Celecoxib for Chronic Uveitis: A Phase I Investigational Safety Study
Brief Title: Intravitreal Celecoxib for Chronic Uveitis
Acronym: Celecoxib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Vanderbilt University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Assistant Professor of Ophthalmology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND for Celecoxib
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Inflammation
Keywords: Macular edema
MeSH Terms: conditions — Inflammation; Macular Edema | interventions — Celecoxib; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib (Experimental): 1-4 mg intravitreal injection ofCelecoxib
  Interventions: Drug: Intravitreal Celecoxib

INTERVENTIONS:
Drug: Intravitreal Celecoxib — 1-4 mg intravitreal celecoxib
  Other Names: Celebrex; NSAIDS

SUMMARY:
Intraocular delivery of celecoxib will be an effective means to treat inflammation and macular edema and prevent structural complications and vision loss in patients with chronic inflammation or macular edema who are unable to tolerate corticosteroids due to their side effects.

DETAILED DESCRIPTION:
Specific Aims I: Test the safety of intraocular injection of 1mg and 4mg celecoxib in patients who have chronic inflammation or macular edema who are unable to tolerate corticosteroids due to their side effects.

II: Test the efficacy of intraocular 1mg and 4mg celecoxib in treating inflammation or structural complications of inflammation (macular edema) in patients who are unable to tolerate corticosteroids due to their side effects.

After investigational new drug application and Vanderbilt Institutional Review Board approval, celecoxib will be compounded by the Investigational Drug Service of the Vanderbilt Medical Center and packaged in individual sterile single use syringes for intraocular injection within 2 hours of preparation. Pharmaceutical grade celecoxib will be obtained from the drug manufacturer (Pfizer) with certificate analysis and compounded in sterile dimethyl sulfoxide following strict sterile technique.

ELIGIBILITY:
Inclusion Criteria:

* Chronic inflammation and/or macular edema despite maximal medical treatment Unable to tolerate corticosteroids due to side effects Aphakic or Pseudophakic subjects

Exclusion Criteria:

* 15 years or younger Have active ocular infection Pregnancy Phakic subjects

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Safety | 12 weeks
  Participant will receive an intravitreal injection of the Celecoxib and be followed for any possible adverse events

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  Participant will receive the intravitreal injection of celecoxib day 1 and be followed for efficacy. The efficacy will be determined from the ophthalmic exams and aqueous samples